CLINICAL TRIAL: NCT01664026
Title: A 6-Month, Randomized Study to Evaluate the Efficacy of a Web-based Lifestyle Modification Program With and Without Telephone Counseling Support
Brief Title: Efficacy of a Web-based Lifestyle Modification Program in Obese Patients With Cardiovascular Risk Factors
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of funds
Sponsor: Clínica Bazterrica (Other)
Responsible Party: Principal Investigator, Arnaldo Angelino, Jefe de Prevencion y Rehabilitacion, Clínica Bazterrica
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PWeb123
Record Dates: First submitted 2012-08-09; First posted 2012-08-14 (Estimated); Last update posted 2019-02-01 (Actual); Status verified 2019-01

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Control (No Intervention): Subjects assigned to the usual care group will receive general lifestyle recommendations as per their country standards of care.
- Web (Experimental): Access to a web-based lifestyle modification program of 6-month duration that covers all aspects of a healthy lifestyle including physical activity, nutrition and weight maintenance.
  Interventions: Behavioral: Web-based lifestyle modification
- Web+ (Experimental): Access to a web-based lifestyle modification program of 6-month duration that covers all aspects of a healthy lifestyle including physical activity, nutrition and weight maintenance plus telephone counseling support by health coaches on a weekly or bi-weekly basis.
  Interventions: Behavioral: Web-based lifestyle modification +

INTERVENTIONS:
Behavioral: Web-based lifestyle modification — Access to a web-based lifestyle modification program of 6-month duration that covers all aspects of a healthy lifestyle including physical activity, nutrition and weight maintenance.
  Arms: Web
Behavioral: Web-based lifestyle modification + — Access to a web-based lifestyle modification program of 6-month duration that covers all aspects of a healthy lifestyle including physical activity, nutrition and weight maintenance plus telephone counseling support by health coaches on a weekly or bi-weekly basis.
  Arms: Web+

SUMMARY:
To evaluate the effect of a 6-month web-based lifestyle modification program with and without telephone counseling versus usual care in obese patients with cardiovascular risk factors on:

* Weight Loss
* Waist circumference; blood pressure; total cholesterol, triglycerides, LDL-cholesterol, HDL-cholesterol; glucose and hemoglobin A1c; C-reactive protein.
* Physical activity and eating habits
* Quality of life

ELIGIBILITY:
Inclusion Criteria:

1. Male or female 25-70 years of age
2. Obese (BMI ≥ 30 kg/m2 and <40 kg/m2)
3. At least 2 cardiovascular risk factors (diabetes, hypertension or dyslipidemia) i) Hypertension defined by a history of hypertension, treatment of hypertension or BP values >140/90 mmHg in two consecutive office visits ii) High cholesterol defined by an LDL-C ≥130 mg/dL and/or HDL-C <40 mg/dL and triglycerides ≥150 mg/dL iii) Type 2 Diabetes Mellitus defined by a history of diabetes, treatment of diabetes or fasting glucose ≥126 mg/dL in two consecutive office visits
4. Participant must be willing and able to provide written informed consent
5. Participant must be willing and able to comply with study related procedures
6. Participant must have access to Internet and e-mail

Exclusion Criteria:

1. Stage 1 or 2 on Patient Activation Measures tool
2. Weight change of more than 5 kg during the 3 months preceding the screening visit
3. History of bariatric surgery
4. Fasting Plasma Glucose at screening > 250 mg/dL (> 13.9 mmol/L)
5. Hemoglobin A1c at screening >8.5%
6. Treatment of type 2 diabetes with insulin (except for history of intermittent acute use, no more than 2 weeks usage in previous 6 months)
7. Uncontrolled or inadequately controlled hypertension at the time of screening with blood pressure >160/100 mmHg
8. Secondary hypertension
9. Changes in lipid, blood pressure or diabetes modifying agents including introduction, change in dose or cessation in the 3 months prior to Screening Visit
10. Personal history of coronary heart disease, congestive heart failure, serious arrhythmias and stroke
11. Cardiovascular, hepatic, neurological, endocrine disease, active malignant tumor or other major systemic disease making implementation of the protocol or interpretation of the study results difficult.
12. Presence of any condition (medical, psychological, social, or geographical), actual or anticipated, that in the opinion of the Investigator would restrict or limit the patient's successful participation for the duration of the study
13. Presence of history of cancer within the past five years with the exception of adequately treated localized basal cell skin cancer or in situ uterine cervical cancer
14. Use of systemic glucocorticoids (excluding topical application or inhaled forms) for one week or more within 3 months prior to the time of screening
15. Use of any investigational agent (drug, biologic, device) within 3 months prior to screening

Ages: 25 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-08; Primary Completion 2013-08 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
Change in body weight from randomization to 6 months | 6 months

SECONDARY OUTCOMES:
Changes in waist circumference | 6 months
Changes in blood pressure | 6 months
Changes in lipid parameters (total cholesterol, triglycerides, LDL-cholesterol, HDL-cholesterol) | 6 months
Changes in glycemic parameters (glucose and hemoglobin A1c) | 6 months
Changes in C-reactive protein | 6 months

OTHER OUTCOMES:
Changes in lifestyle behaviors (physical activity and eating habits) | 6 months
Changes in quality of life | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Andres Digenio, MD, Study Director
Locations (1):
- Clinica Bazterrica, Buenos Aires, Argentina